CLINICAL TRIAL: NCT05366309
Title: OUtcome Following Tailored Education and Retraining: Studying Performance and Adherence in ChildrEn and Young People With Asthma: a Randomised Feasibility Study
Brief Title: Performance and Adherence in Children Using Spacers
Acronym: OUTER-SPACERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3022
Record Dates: First submitted 2022-04-20; First posted 2022-05-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Asthma; Asthma in Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Control) Group (Active Comparator): Participants randomised to this group will receive usual care in terms of their education.
  Interventions: Other: Standard care education
- Tailored Education Group (Experimental): Participants randomised to this group will receive tailored education, which is additional to standard care.
  Interventions: Other: Tailored education

INTERVENTIONS:
Other: Tailored education — Tailored Education: A delegated investigator will review the SD memory card data and share the results with the participant and/or parent/guardian. The investigator will explain whether there are partial or critical errors to inhalation technique that have been recorded. The participant will be informed about their overall adherence; including how and when they used their asthma medications. If errors in medication use are identified, specific coaching will be provided to help eliminate errors.
  Arms: Tailored Education Group
Other: Standard care education — Participants randomised to this group will receive usual care in terms of their education.
  Arms: Standard Care (Control) Group

SUMMARY:
Asthma is a common disease which causes swelling in the airways, making it difficult to breathe. Asthma is common in children, affecting 1 in 11 children in the UK. Asthma is treated with inhalers which reduce the swelling. If inhalers are taken correctly they can help keep symptoms under control, allowing asthma sufferers to go about their day with less chance of having an asthma attack. Many patients have been found to not take their inhalers correctly and either under use (which leads to poor control of symptoms) or over use (which leads to potential side effects).

Although asthma in most patients can be controlled with inhalers, not using inhalers correctly is one of the most common causes of poor control. This is common in children and young people (CYP) with all severities of asthma, resulting in high burden on the families and healthcare systems.

The biggest challenge facing doctors and nurses helping CYP with asthma is finding a way to ensure that they take the medication. Whilst there are many studies looking into inhaler use, there are no large studies about how inhalers are used between clinic visits in CYP with asthma.

The Smart Spacer is monitoring device which allows doctors to monitor when and how effectively inhalers are being used. This study wants to find out how well this device works, how well and how often CYP are using their inhalers, and if tailored education improves asthma control. To do this, participants in the study will be randomly selected to have "tailored education" or "standard care education".

The investigators are inviting 100 children and young people (CYP) aged 6-18 years who have asthma to join this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-18 years;
* Attending secondary care with a diagnosis of asthma;
* Willing and able to give fully informed consent, or, participants having an acceptable individual capable of giving consent on the participant's behalf (e.g. parent or guardian of a child under 16 years of age);
* Able to perform lung function and exhaled nitric oxide measurements;
* Take twice-daily preventer medication using a valved holding chamber (spacer device) i.e. inhaled corticosteroid with or without long-acting beta antagonist;
* Willing and able to comply with the study procedures.

Exclusion Criteria:

* Significant co-existing respiratory disease (e.g. cystic fibrosis);
* Currently participating in another clinical trial of an investigational medicinal product or medical device;
* Non-English speaker where translation facilities are insufficient to guarantee informed consent.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall adherence to inhaled treatment (the product of persistence (number of doses taken as prescribed) and technique) | From recruitment up until 12-16 weeks follow-up time point
  Overall adherence

SECONDARY OUTCOMES:
The proportion of children and young people with asthma who are eligible for participation within the study from secondary care via screening logs | From recruitment up until 12-16 weeks follow-up time point
  Proportion eligible
Recruitment and attrition rates over the study via screening and enrolment logs | From recruitment up until 12-16 weeks follow-up time point
  Recruitment and attrition
The success rate of obtaining data from the Smart spacer device | From recruitment up until 12-16 weeks follow-up time point
  Success rate
Feedback from System Usability Score (SUS) | At 12-16 weeks follow-up time point
  SUS
Feedback from Net Promoter Score (NPS) | At 12-16 weeks follow-up time point
  NPS
Rate of device failure from any cause (including loss of device, inability to retrieve data from SD card) | From recruitment to 12-16 weeks follow-up time point
  Device failure
Asthma control test (ACT) or Childhood Asthma Control Test (c-ACT) | From recruitment to 12-16 weeks follow-up time point
  ACT
Asthma Control Questionnaire | From recruitment to 12-16 weeks follow-up time point
  ACQ
GINA control score | From recruitment to 12-16 weeks follow-up time point
  GINA
Salbutamol (rescue) use | From recruitment to 12-16 weeks follow-up time point
  Salbutamol use
Need for oral steroid burst | From recruitment to 12-16 weeks follow-up time point
  Oral steroid burst use
m-PAQLQ score | From recruitment to 12-16 weeks follow-up time point
  m-PAQLQ
FEV1 z score | From recruitment to 12-16 weeks follow-up time point
  FEV1 z
FeNO (ppb) | From recruitment to 12-16 weeks follow-up time point
  FeNO (ppb)
UKIG score | From recruitment to 12-16 weeks follow-up time point
  UKIG

CONTACTS AND LOCATIONS:
Overall Officials: Will Carroll, Principal Investigator — PI
Locations (1):
- Robert James Bowler, Stoke-on-Trent, Staffordshire, United Kingdom